# **S1929** Research Study Informed Consent Document (Treatment Study Consent)

**Study Title for Participants:** Testing Maintenance Therapy for Small Cell Lung Cancer in Patients with SLFN11 Positive Biomarker

# Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>:

<u>S1929</u>, "Phase II Randomized Study of Maintenance Atezolizumab versus Atezolizumab in Combination with Talazoparib in Patients with SLFN11 Positive Extensive Stage Small Cell Lung Cancer (ES-SCLC)" NCT#: 04334941

# Overview and Key Information (This section is a summary of the treatment consent form)

# What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have extensive stage small cell lung cancer (ES-SCLC) and have been tested SLFN11 positive.

# Taking part in this study is your choice.

You can choose to take part, or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.



# Why is this study being done?

This study is being done to answer the following question:

Can we lower the chance of small cell lung cancer growing or spreading by adding talazoparib to the usual atezolizumab treatment?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for small cell lung cancer. The usual approach is defined as care most people get for small cell lung cancer.

# What is the usual approach to treating my small cell lung cancer?

The usual approach for patients who are not in a study is treatment with atezolizumab alone.

# What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

# What will happen if I decide to take part in this treatment study?

If you are eligible and decide to take part in this study, you will either get the study drugs atezolizumab and talazoparib, or you will get atezolizumab alone.

After you finish your treatment, your doctor and study team will watch you for side effects. They will check you every 6 months for 2 years and at the end of Year 3 from the start of treatment. This means you will keep seeing your doctor for up to 3 years from the time you start treatment.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.



#### **Risks**

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that adding talazoparib may not be as good as taking atezolizumab alone at stabilizing the cancer.

There is also a risk that you could have side effects from the study drugs. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:

- Anemia, tiredness
- Headache
- Hair loss
- Decreased appetite
- Shortness of breath
- Nausea, vomiting, diarrhea
- Bruising, bleeding
- Infection, especially when white blood cell count is low

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is evidence that the study approach is effective in stabilizing your type of cancer. It is not possible to know now if the study drugs will extend your time without disease compared to the usual approach. This study will help the study doctors learn things that will help people in the future.

# If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. This may mean slowly stopping the study drugs so that there is not a sudden unsafe dosing change that might put your health at risk. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

# Are there other reasons why I might stop being in the study?



Yes. The study doctor may take you off the study if:

- Your health changes and the study are no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (SWOG). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

# What is the purpose of the treatment study?

The purpose of the treatment study is to compare the usual treatment (atezolizumab) alone to using talazoparib plus the usual treatment. The addition of talazoparib to the usual treatment could prevent cancer from growing, but it could also cause side effects, which are described in the risks section below.

This study will help the study doctors find out if this different approach is better than the usual approach. To decide if it is better, the study doctors will be looking to see if the atezolizumab and talazoparib will stabilize the cancer compared to the usual approach.

This immunotherapy drug, atezolizumab, is already approved by the FDA for use in ES-SCLC cancer. There will be about 94 people taking part in this study.

# What are the study groups?

If the tumor is SLFN11 positive and you meet all other study requirements, then you will be randomized to a study group.



This study has 2 study groups.

#### • Group 1

If you are in this group, you will be given atezolizumab through a vein in the arm over 60 minutes, followed by a 30-minute observation time, once every 21 days. This drug is approved by the FDA.

There will be about 47 people in this group.

#### • Group 2

If you are in this group, you will get talazoparib plus atezolizumab. You will take talazoparib by mouth once a day, at around the same time each day (preferably in the morning). It is important to swallow whole and not to chew the capsules. Talazoparib can be taken with or without food. Always use gloves when handling talazoparib capsules. You will be given atezolizumab through a vein in the arm over 60 minutes, followed by a 30-minute observation time, once every 21 days.

You also will keep a pill diary. This helps you keep track of when you take your pills. The study doctor will show you how to use this diary. Each time you visit the clinic, you must bring the pill diary, any remaining pills, and the pill bottle.

There will be about 47 people in this group.

We will use a computer to assign you to one of the study groups. This process is called "randomization." It means that your doctor will not choose, and you cannot choose which study group you are in. You will be put into a group by chance. You will have an equal chance of being in Group 1 or Group 2.



Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right following the lines and arrows.



# What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Some exams, tests, and procedures are a necessary part of the research study but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

SLFN11 testing
 This testing is done during the screening step of this study and is discussed in the screening consent.

Your study doctor will need to use some of the tissue left over from your biopsy when you were diagnosed with cancer. This is discussed in the screening consent.

You will be given the option to store additional tissue in the biobank. Storing samples is called "biobanking" and the biobank is run by SWOG and is supported by the NCI. This will be discussed in the section under "Optional studies" below.



# What risks can I expect from taking part in the treatment study?

#### **General Risks**

you choose to take part in this study, there is a risk that the study approach may not be as good as the usual approach for your cancer at stabilizing your cancer. You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The drugs used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 5 months after you have completed the study.

#### **Side Effect Risks**

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drugs.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.



S1929 Treatment Consent Page 8 Version Date 11/18/2024

This study is looking at a combination of the usual drugs used to treat this type of cancer plus a study drug. This different combination of drugs may increase your side effects or may cause new side effects.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

#### Possible Side Effects of Atezolizumab

(CAEPR Version 2.4, September 14,2023)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving atezolizumab (MPDL3280A), more than 20 and up to 100 may have:

- Tiredness
- Infection



#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving atezolizumab (MPDL3280A), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Diarrhea, nausea, vomiting
- Difficulty swallowing
- Fever
- Flu-like symptoms including body aches
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Reaction during or following a drug infusion which may cause fever, chills, rash
- Loss of appetite
- Pain in back
- Cough, shortness of breath, stuffy nose
- Itching, acne, rash

Atezolizumab (MPDL3280A) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches, extreme tiredness or changes in mood or behavior decreased sex drive; weight loss or weight gain; excessive thirst or urine; dizziness or fainting.
- Pain in belly
- Pain or swelling of the joints
- Rash that develops on skin, nails, scalp and inside of mouth or vagina that may be painful



#### RARE, AND SERIOUS

In 100 people receiving atezolizumab (MPDL3280A), 3 or fewer may have:

Bruising, bleeding

Atezolizumab (MPDL3280A) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Heart problems including swelling and heart failure. Symptoms and signs of heart problems may include: shortness of breath, swelling of the ankles and body.
- A condition with high blood sugar which leads to tiredness, frequent urination or excessive thirst
- Swelling and redness of the eye
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine. Signs and symptoms of colitis may include: diarrhea or increase in bowel movements, blood in your stools or dark, tarry, sticky stools, severe belly pain or tenderness.
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting; drowsiness; pain in the right upper belly.
- Damage to organs in the body when the body produces too many white cells
- Swelling of the brain (meningitis/encephalitis), which may cause: headache, confusion, sleepiness, seizures, and stiff neck
- Abnormal movement of the facial muscles
- Swelling of the spinal cord
- Problem of the muscle, including swelling, which can cause muscle pain and severe muscle weakness sometimes with dark urine
- Problem of the nerves that can cause paralysis. Signs and symptoms may include: numbness, tingling of hands and feet; weakness of the arms, legs.
- Kidney problems, including nephritis and kidney failure requiring dialysis. Signs of kidney problems may include: decrease in the amount of urine, blood in your urine, ankle swelling.
- Lung problems (pneumonitis and pleural effusion). Symptoms may include: new or worsening cough, chest pain, shortness of breath.
- Skin: blisters on the skin, including inside the mouth (can be severe), rash with blisters, skin rash developing 1-8 weeks after a drug is given, which may be accompanied by fever, lymph node swelling and organ failure.



#### Possible Side Effects of Talazoparib

(CAEPR Version 2.5: September 23, 2024)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving talazoparib (PF-06944076), more than 20 and up to 100 may have:

- Anemia which may require blood transfusion
- Nausea
- Tiredness
- Bruising, bleeding
- Loss of appetite

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving talazoparib (PF-06944076), from 4 to 20 may have:

- Pain
- Constipation, diarrhea, heartburn, vomiting
- Sores in the mouth which may cause difficulty swallowing
- Fever
- Infection, especially when white blood cell count is low
- Dizziness, headache
- Changes in taste
- Hair loss

#### RARE, AND SERIOUS

In 100 people receiving talazoparib (PF-06944076), 3 or fewer may have:

- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require transfusions
- A new cancer resulting from treatment of earlier cancer

#### **Additional Drug Risks**

#### **Drug Interactions**

The study drug could interact with other drugs and herbal medicines.

Over the counter, herbal medicines and other prescribed drugs will be reviewed by the study team for potential drug interactions. Your doctor or a member of the study team will tell you if you need to stop, modify or change any of these medicines or drugs before you start taking talazoparib and atezolizumab.

Any medications or substances that contain strong P-gp or BCRP inhibitors should be avoided while you are taking talazoparib. Caution should be used for coadministration of other P-gp inhibitors (e.g., amiodarone, azithromycin, captopril, carvedilol, clarithromycin, conivaptan, cyclosporine, diltiazem, erythromycin, felodipine, lopinavir, quercetin), P-gp inducers (e.g., avasimibe, carbamazepine, phenytoin, St John's wort), or BCRP inhibitors (e.g., cyclosporine, eltrombopag, and gefitinib).



Throughout your treatment, you should inform your doctor about any medication changes.

Do not receive any live attenuated vaccinations, such as shingles or influenza nasal spray, while you are taking part in this study.

Rarely, there are problems getting enough supplies of the study drugs. If that happens, your doctor will talk with you about your options.

Your study doctor will give you a drug information handout and wallet card that lists these possible interactions. Share this information with your family members, caregivers, other health care providers, and pharmacists

# What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.
- Write down in your medication diary when you take the study drug at home.

**For women:** Do not get pregnant or breastfeed while taking part in this study. **For men:** Do not father a baby while taking part in this study. Do not donate sperm while taking part in this study and for 4 months after your last dose of the study drugs. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 7 months after your last dose of the study drugs.

# What are the costs of taking part in the treatment study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your small cell lung cancer. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the costs of getting talazoparib and atezolizumab ready and giving it to you.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.



S1929 Treatment Consent Page 13 Version Date 11/18/2024

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You or your insurance provider will not have to pay for talazoparib and atezolizumab while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What happens if I am injured because I took part in the treatment study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.



### Some of these organizations are:

- The study sponsor, SWOG, and any company supporting the study now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

# Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).



S1929 Treatment Consent Page 15 Version Date 11/18/2024

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

| You can talk to the study doctor report side effects or injuries. C | about any questions or concerns you have contact the study doctor | e about this study or to (insert name of |
|---|---|---|
| study doctor[s]) at | | \ |
| For questions about your rights | while in this study, call the | (insert name |
| of organization or center) Instit<br>number). | utional Review Board at | (insert telephone |

# Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the treatment study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people with cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the treatment study even if you say "no" to any or all of these studies. There is no penalty for saying "no." You and your insurance company will not be billed for these optional studies. If you sign up for but cannot complete any of these studies for any reason, you can still take part in the treatment study.

Circle your choice of "yes" or "no" for each of the following studies.

# Optional sample collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

#### Unknown future studies

If you choose to take part in this optional study, your blood and tissue samples will be collected and stored. Storing samples for future studies is called "biobanking." The biobank is being run by SWOG and is supported by the NCI. This is a publicly funded study. Samples from publicly



funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we don't know what research may be done in the future using your blood and tissue samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes. If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal tissue and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.

#### What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

- 1. Less than 3 teaspoons of blood will be collected from a vein in your arm at cycles 1, 3, and every 12 weeks until your disease gets worse or you stop treatment.
- 2. A sample from the tissue that was already removed by surgery or biopsy, will be sent to the biobank.
- 3. Your sample will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 4. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 5. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

#### What are the risks in this optional sample collection?



- The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: https://www.genome.gov/10002328/

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your sample and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.



#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

#### What if I change my mind about this optional sample collection?

| If you decide you no longer want your samples to be used, you can call the study doctor, (insert name of study doctor for main trial) at |
|---|
| (insert telephone number of study doctor for main trial), who will let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers. |
| What if I have questions about this optional sample collection? |
| If you have questions about the use of your samples for research, contact the study doctor, (insert name of study doctor for main trial) at |
| (insert telephone number of study doctor for main trial). |
| Please circle your answer below to show if you would or would not like to take part in each optional study: |
| Samples for unknown future studies: |

health research.

YES

### **Contact for Future Research**

NO

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

I agree that my samples and related health information may be kept in a biobank for use in future

| YES | NO |
|-----|----|



# This is the end of the section about optional studies.

My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree

to take part in the treatment study. I also agree to take part in any additional studies where I circled "yes".

| Participant's signature (or legally authorized representative) |
|-------------------------------------------------------------------|
| Date of signature |
| Signature of person(s) conducting the informed consent discussion |
| Date of signature |

